CLINICAL TRIAL: NCT01198574
Title: The Role of Sub-clinical Inflammation on the Iron Status of Myanmar Anaemic Adolescent Schoolgirls During Iron and Vitamin A Supplementation
Brief Title: Sub-clinical Inflammation and Iron Supplementation
Acronym: SCI&Anaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Department of Medical Research, Lower Myanmar (Other)
Responsible Party: Principal Investigator, Min Kyaw Htet, Dr, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCIVA
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Results first posted 2012-05-16 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Anemia
Keywords: anemia; iron supplementation; sub-clinical inflammation; adolescents
MeSH Terms: conditions — Anemia | interventions — Iron-Dextran Complex; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Iron group (Experimental)
  Interventions: Dietary Supplement: Iron group
- Vitamin A group (Experimental): Vitamin A group
  Interventions: Dietary Supplement: Vitamin A group
- Iron and Vitamin A group (Experimental): Iron and Vitamin A group
  Interventions: Dietary Supplement: Iron and vitamin A group
- Placebo group (Experimental): Placebo group with folic acid
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Iron group — Ferrous fumarate, 60 mg, weekly dose
  Other Names: Iron supplement
  Arms: Iron group
Dietary Supplement: Vitamin A group — Retinol, weekly dose, 15,000 IU
  Other Names: Vitamin A supplement
  Arms: Vitamin A group
Dietary Supplement: Iron and vitamin A group — Ferrous fumarate, Retinol combination group, weekly dose
  Other Names: Iron and Vitamin A supplement
  Arms: Iron and Vitamin A group
Dietary Supplement: Placebo group — folic acid only as placebo group
  Other Names: Placebo group, folic acid only
  Arms: Placebo group

SUMMARY:
Anemia and vitamin A deficiency (VAD) are major nutritional problems in the world and also in Myanmar. Both nutrient deficiencies result from interaction of several causal factors, and a better understanding of the etiology to interpret the prevalence and to formulate appropriate measures to reduce these deficiencies is necessary. There is a growing concern on the role of sub-clinical inflammation on the nutritional status indicators during the nutritional status assessment. However, there is lack of information on the role of inflammation on the iron supplementation. The adolescent period is a window of opportunity to improve the preconceptional iron status of the girls and recently gained much attention. The purpose of the study is to understand the role of inflammation on iron and vitamin A status during iron and vitamin A supplementation. The findings will show the extent to which iron supplementation has been hampered by inflammation and to formulate the necessary measures to overcome the interference.

ELIGIBILITY:
Inclusion Criteria:

* adolescent girls (age 12-19 years)
* already experienced menarche
* anemic girls (Hb<120 g/L)
* no known illness (apparently healthy)
* free from haemoglobinopathy
* No regular consumption of iron and vitamin A supplement during the last 3 months

Exclusion Criteria:

* subjects with chronic illness
* subjects with severe anaemia
* who do not give the consents

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 402 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyaw Htet, PhD, Principal Investigator — (1) South East Asian Ministers of Education Organization, Regional Center for Food and Nutrition, University of Indonesia, (2) Ministry of Health, Myanmar
Locations (1):
- Nyaung Done Township, Pathein, Ayeyarwady Region, Burma

REFERENCES:
- [Background] Thurnham DI, McCabe LD, Haldar S, Wieringa FT, Northrop-Clewes CA, McCabe GP. Adjusting plasma ferritin concentrations to remove the effects of subclinical inflammation in the assessment of iron deficiency: a meta-analysis. Am J Clin Nutr. 2010 Sep;92(3):546-55. doi: 10.3945/ajcn.2010.29284. Epub 2010 Jul 7. PMID 20610634
- [Background] Mburu AS, Thurnham DI, Mwaniki DL, Muniu EM, Alumasa F, de Wagt A. The influence and benefits of controlling for inflammation on plasma ferritin and hemoglobin responses following a multi-micronutrient supplement in apparently healthy, HIV+ Kenyan adults. J Nutr. 2008 Mar;138(3):613-9. doi: 10.1093/jn/138.3.613. PMID 18287375
- [Background] Thurnham DI, Mburu AS, Mwaniki DL, Muniu EM, Alumasa F, de Wagt A. Using plasma acute-phase protein concentrations to interpret nutritional biomarkers in apparently healthy HIV-1-seropositive Kenyan adults. Br J Nutr. 2008 Jul;100(1):174-82. doi: 10.1017/S0007114507883012. Epub 2008 Jan 4. PMID 18177514
- [Background] Thurnham DI, Mburu AS, Mwaniki DL, De Wagt A. Micronutrients in childhood and the influence of subclinical inflammation. Proc Nutr Soc. 2005 Nov;64(4):502-9. doi: 10.1079/pns2005468. PMID 16313694
- [Background] Thurnham DI. Vitamin A, iron, and haemopoiesis. Lancet. 1993 Nov 27;342(8883):1312-3. doi: 10.1016/0140-6736(93)92239-p. No abstract available. PMID 7901629
- [Background] Angeles-Agdeppa I, Schultink W, Sastroamidjojo S, Gross R, Karyadi D. Weekly micronutrient supplementation to build iron stores in female Indonesian adolescents. Am J Clin Nutr. 1997 Jul;66(1):177-83. doi: 10.1093/ajcn/66.1.177. PMID 9209187
- [Background] Tee ES, Kandiah M, Awin N, Chong SM, Satgunasingam N, Kamarudin L, Milani S, Dugdale AE, Viteri FE. School-administered weekly iron-folate supplements improve hemoglobin and ferritin concentrations in Malaysian adolescent girls. Am J Clin Nutr. 1999 Jun;69(6):1249-56. doi: 10.1093/ajcn/69.6.1249. PMID 10357747
- [Derived] Htet MK, Fahmida U, Dillon D, Akib A, Utomo B, Thurnham DI. The influence of vitamin A status on iron-deficiency anaemia in anaemic adolescent schoolgirls in Myanmar. Public Health Nutr. 2014 Oct;17(10):2325-32. doi: 10.1017/S1368980013002723. Epub 2013 Oct 16. PMID 24128336
- [Derived] Htet MK, Dillon D, Akib A, Utomo B, Fahmida U, Thurnham DI. Microcytic anaemia predominates in adolescent school girls in the delta region of Myanmar. Asia Pac J Clin Nutr. 2012;21(3):411-5. PMID 22705432
- See also: South East Asian Ministers of Education Organization, Regional Center for Food and Nutrition, University of Indonesia — http://www.seameo-recfon.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening for the study subjects was conducted in July, 2010 among the adolescent schoolgirls in Nyaung Done Township, Irrawaddy Division. It included assessment of Hb status using the Coulter Counter. Information on the general characteristics and menarche status of the girls are obtained.
Pre-assignment Details: Deworming with 400 mg Albendazole was done one week before the baseline data collection.
Groups:
- Iron Group: Iron group received 60 mg of elemental iron, 2.5 mg folic acid + Placebo Vitamin A weekly
- Vitamin A Group: Vitamin A group received 15,000 IU Vitamin A + Placebo iron containing 2.5 mg folic acid weekly
- Iron and Vitamin A Group: Iron and Vitamin A group received 60 mg elemental iron, 2.5 mg folic acid + 15,000 IU Vitamin A weekly
- Placebo Group: Placebo group received 2.5 mg folic acid weekly
Period: Overall Study
Arm/Group | Iron Group | Vitamin A Group | Iron and Vitamin A Group | Placebo Group
Started | 98 | 102 | 100 | 102
Completed | 94 | 101 | 99 | 98
Not Completed | 4 | 1 | 1 | 4
Not completed — Resigned from schools | 4 | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Iron Group: Iron group received 60 mg elemental iron, 2.5 mg folic acid with vitamin A placebo weekly
- Vitamin A Group: Vitamin A group received 15,000 IU Vitamin A + Iron placebo with 2.5 mg folic acid weekly
- Iron and Vitamin A Group: Iron and Vitamin A group received 60 mg elemental iron, 2.5 mg folic acid +15,000 IU Vitamin A weekly
- Placebo Group: Placebo group received iron placebo containing 2.5 mg folic acid weekly
- Total: Total of all reporting groups
Arm/Group | Iron Group | Vitamin A Group | Iron and Vitamin A Group | Placebo Group | Total
Number analyzed (Participants) | 98 | 102 | 100 | 102 | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 98 | 102 | 100 | 102 | 402
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 15.9 (1.2) | 16.1 (1.2) | 16.1 (1.2) | 15.8 (1.1) | 16.0 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 102 | 100 | 102 | 402
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Myanmar | 98 | 102 | 100 | 102 | 402

OUTCOME MEASURES:

1. Primary Outcome: Haemoglobin Level
Description: Haemoglobin level (g/L) measured by cyanmethaemoglobin method
Time Frame: at week 0, week 6 and week12
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Iron Group: 60 mg Elemental iron with 2.5 mg folic acid + Vitamin A placebo
- Vitamin A Group: 15,000 IU vitamin A + Iron Placebo containing 2.5 mg folic acid
- Iron and Vitamin A Group: 60 mg Elemental iron with 2.5 mg folic acid + Vitamin A 15,000 IU
- Placebo Group: 2.5 mg folic acid + Vitamin A placebo
Arm/Group | Iron Group | Vitamin A Group | Iron and Vitamin A Group | Placebo Group
Number analyzed (Participants) | 94 | 101 | 98 | 98
g/L
  Hb week 0 (Baseline) | 88.3 (11.2) | 89.2 (11.5) | 88.4 (12.1) | 89.6 (12.7)
  Hb week 6 (Midline) | 98.1 (10.6) | 98.7 (9.6) | 99.2 (10.0) | 98.3 (10.7)
  Hb week 12 (Endline) | 110.8 (9.8) | 109.0 (9.1) | 111.4 (9.0) | 109.7 (8.4)
Statistical Analysis 1: Comparison: Iron Group vs Vitamin A Group vs Iron and Vitamin A Group vs Placebo Group; Null Hypothesis 1. Haemoglobin level was not influenced by sub-clinical inflammation during iron supplementation in the anaemic adolescent school girls 2. Vitamin A does not improve the haemoglobin level of the anaemic schoolgirls during iron supplementation in the presence of inflammation; Test type: Superiority or Other; p < 0.05, GLM for repeated measures; The Hb concentration at Week 0, Week 6 and Week 12 are analyzed using GLM repeated measures

2. Primary Outcome: Status of Tissue Iron Store
Description: Tissue iron store was measured by serum ferritin
Time Frame: at week 0, week 6 and week12
Population: Per Protocol analysis
Measure: Geometric Mean (Standard Deviation); unit: µg/L
Arm/Group | Iron Group | Vitamin A Group | Iron and Vitamin A Group | Placebo Group
Number analyzed (Participants) | 94 | 101 | 98 | 98
µg/L
  serum ferritin (Baseline) | 32.1 (2.5) | 34.4 (2.6) | 25.9 (3.1) | 31.1 (2.5)
  serum ferritin (Midline) | 34.5 (1.9) | 32.1 (2.3) | 32.3 (2.1) | 26.5 (2.3)
  serum ferritin (Endline) | 39.6 (2.1) | 35.0 (2.5) | 35.4 (2.4) | 28.2 (2.5)
Statistical Analysis 1: Comparison: Iron Group vs Vitamin A Group vs Iron and Vitamin A Group vs Placebo Group; Null hypothesis 1. Iron status indicator (serum ferritin) was not influenced by sub-clinical inflammation during iron supplementation in the anaemic adolescent school girls 2. Vitamin A does not improve the iron status indicator (serum ferritin) concentration of the anaemic schoolgirls during iron supplementation in the presence of inflammation; Test type: Superiority or Other; p < 0.05, GLM for repeated measures ANOVA

3. Primary Outcome: Status of Cellular Iron Deficiency
Description: Cellular Iron deficiency status is also measured by serum transferrin receptor
Time Frame: at week 0, week 6 and week12
Population: Per Protocol analysis
Measure: Geometric Mean (Standard Deviation); unit: mg/L
Arm/Group | Iron Group | Vitamin A Group | Iron and Vitamin A Group | Placebo Group
Number analyzed (Participants) | 94 | 101 | 98 | 98
mg/L
  serum transferrin receptor (Baseline) | 7.09 (1.52) | 6.56 (1.42) | 7.16 (1.59) | 6.74 (1.50)
  serum transferrin receptor (Midline) | 6.69 (1.51) | 6.39 (1.41) | 6.73 (1.53) | 6.59 (1.53)
  serum transferrin receptor (Endline) | 6.44 (1.55) | 6.27 (1.44) | 6.24 (1.43) | 6.61 (1.54)
Statistical Analysis 1: Comparison: Iron Group vs Vitamin A Group vs Iron and Vitamin A Group vs Placebo Group; Null Hypothesis 1. iron status indicator (sTfR) was not influenced by sub-clinical inflammation during iron supplementation in the anaemic adolescent school girls 2. Vitamin A does not improve iron status indicator (sTfR) of the anaemic schoolgirls during iron supplementation in the presence of inflammation; Test type: Superiority or Other; p < 0.05, GLM for repeated measures ANOVA

ADVERSE EVENTS:
Time Frame: The adverse effect of supplementation were collected weekly throughout the 12 weeks of intervention.
Arm/Group | Iron Group | Vitamin A Group | Iron and Vitamin A Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/102 | 0/100 | 0/102
Other Adverse Events (participants affected / at risk) | 0/98 | 0/102 | 0/100 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No